CLINICAL TRIAL: NCT05524909
Title: Combined Effects of Communicating Genetic Risk of Type 2 Diabetes and Wearable Technologies on Objectively Measured Behavioral Outcomes in Overweight or Obese East Asian Individuals.
Brief Title: Full-scale Intervention Study: Genetic Risk Communication and Wearables
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kim, Youngwon, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: geneticriskwearabletrial_full
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Fitness Trackers; Physical Activity; Exercise; Genetic Predisposition to Disease; Type 2 Diabetes
Keywords: type 2 diabetes; physical activity; genetic risk; wearable technology; randomized controlled trial; movement behavior; nutrition
MeSH Terms: conditions — Motor Activity; Genetic Predisposition to Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: parallel-group, open randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Group allocation will be concealed from study staff until the 7-day pre-intervention period begins (for preparation of corresponding e-leaflets, genetic risk estimates and/or baseline Fitbit step goal calculations), and from participants until the interventions are delivered. Given the nature of the interventions delivered, it will be impossible for participants to be blinded to the specific intervention they receive once the initial interventions are provided; however, study staff analyzing participants' de-identified data will remain blinded to participant randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): The control group will receive a Fitbit device
- Intervention Group - Genetic Risk Estimate (Experimental): This intervention group will receive an estimated genetic risk and e-leaflet of type 2 diabetes in addition to the Fitbit .
  Interventions: Genetic: Genetic Risk Estimate
- Intervention Group - Genetic Risk Estimate + Fitbit Functions (Experimental): This intervention group will receive a Fitbit device, but have a Fitbit step goal set 10% higher than their baseline step count, and use its prompt functions, in addition to the genetic risk estimate and e-leaflet.
  Interventions: Device: Genetic Risk Estimate + Fitbit Functions

INTERVENTIONS:
Genetic: Genetic Risk Estimate — The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for T2D as well as a dichotomized genetic risk category: 'increased genetic risk' (if their genetic risk is higher than the average population risk) or 'no increased genetic risk' (if their genetic risk is not higher than the average population risk).
  Arms: Intervention Group - Genetic Risk Estimate
Device: Genetic Risk Estimate + Fitbit Functions — The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for T2D as well as a dichotomized genetic risk category: 'increased genetic risk' (if their genetic risk is higher than the average population risk) or 'no increased genetic risk' (if their genetic risk is not higher than the average population risk).
  The two unique Fitbit functions are step goal setting and prompts. Individualized daily step goals will be set to be 10% higher than participants' own baseline Fitbit step counts. The 'Reminder To Move' function of Fitbit will be used as a prompt to remind participants to reduce sedentary time and walk at least 250 steps/hour within a specified timeframe (i.e., from 9am to 10pm in the proposed research). If the user has not accumulated at least 250 steps/hour, a reminder (for example, 150 steps to go) will appear on the Fitbit screen at 10 minutes before the hour (for example, at 10:50 a.m.) and cause the device to vibrate.
  Arms: Intervention Group - Genetic Risk Estimate + Fitbit Functions

SUMMARY:
Background: Communication of information about risk of type 2 diabetes (T2D) alone has not been associated with changes in habitual behaviors among individuals of European ancestry. In contrast, the use of wearable devices that monitor physical activity (PA) has been associated with changes in behavior in some studies. It is uncertain whether risk communication might enhance the effects of wearable devices. We aim to assess the effects on wearable-device-measured PA of communicating genetic risk for T2D alone or in combination with goal setting and activity prompts from a wearable device among overweight or obese East Asians.

Methods: In a parallel group, randomized controlled trial, a total of 355 overweight or obese East Asian individuals aged 40-60 years will be allocated into one of three groups: 1 control and 2 intervention groups. Blood samples will be used for estimation of T2D genetic risk and analysis of metabolic risk markers. Genetic risk of T2D will be estimated based on 113 SNPs associated with T2D among East Asians using an established method. All three groups will receive a Fitbit device. Both intervention groups will be given T2D genetic risk estimates along with lifestyle advice, but one of the intervention groups will additionally use Fitbit's step-goal setting and prompt functions. Questionnaires and physical measurements will be administered at baseline, immediately after intervention delivery, and 6 and 12-month post-intervention following standard operating procedures. The primary outcome is time spent in moderate-to-vigorous PA measured through the Fitbit. Secondary outcomes include other parameters of wearable-device-measured PA, sedentary time, and sleep, body mass index, systolic and diastolic blood pressure, five intermediate metabolic risk markers, hand grip strength, self-reported PA, self-reported fruit and vegetable consumption and smoking status, and a list of psychological variables.

Discussion: This study will be the first randomized controlled trial using the combination of communication of T2D genetic risk with standard functions of wearable devices in any population. Findings will inform strategies to prevent T2D through lifestyle modification.

ELIGIBILITY:
Inclusion Criteria:

* East Asian ancestry
* Aged 40-60 years
* overweight or obese (i.e. measured BMI ≥23 kilograms/meters2 according to the WHO BMI-defined cut-offs for Asians)
* Able to perform daily-living physical activity
* using English/Chinese and a smartphone in Hong Kong

Exclusion Criteria:

* have been diagnosed with any type of diabetes
* pregnant or lactating
* unable to perform daily-life physical activities (determined through Physical activity Readiness Questionnaire [PAR-Q])
* participating in another research study or exercise programs
* had experience of genetic testing
* and/or cannot comprehend English/Chinese (i.e., sole language medium for the study).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 355 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Moderate to Vigorous Physical Activity Minutes between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, 12-month post-intervention, 6-month follow-up
  Moderate to Vigorous Physical Activity Minutes (per day) will be objectively measured by the Fitbit tracker.

SECONDARY OUTCOMES:
Changes in body mass index (BMI) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Measured height (in meters) and body weight (in kilograms) will be combined to report BMI in kg/m^2
Changes in systolic blood pressure between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Systolic blood pressure (mm Hg) will be measured using the OMRON HEM-907 Digital Automatic Blood Pressure Monitor.
Changes in diastolic blood pressure between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Diastolic blood pressure (mm Hg) will be measured using the OMRON HEM-907 Digital Automatic Blood Pressure Monitor.
Changes in hand grip strength between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Hand grip strength (in kilograms) will be measured using the Jamar Hydraulic Hand Dynamometer, which has good reliability and reproducibility.
Changes in Hemoglobin A1c (HbA1c) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including HbA1c (%).
Changes in Total cholesterol between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including Total cholesterol (mmol/L).
Changes in High-density lipoproteins (HDL) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including HDL (mmol/L).
Changes in Low-density lipoproteins (LDL) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including LDL (mmol/L).
Changes in Triglycerides between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including Triglycerides (mmol/L).
Changes in Self-reported Physical Activity between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Fruit and Vegetable Consumption between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Smoking Status between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Psychological Status between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in five activity indicators (steps, 'sedentary minutes', 'lightly active minutes', calories burn, and sleep time) | Baseline, 12-month post-intervention, 6-month follow-up
  steps, sedentary minutes, lightly active minutes, calories burn, and sleep time will be objectively measured by the Fitbit tracker.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Lab, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The datasets analysed during the current study and statistical code are available from the corresponding author on reasonable request, as is the full protocol.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The datasets analysed during the current study and statistical code will be available after the completion of the study
Access Criteria: IPD data can be accessed based on reasonable request by contacting the corresponding author.

REFERENCES:
- [Derived] Ho HHS, Chen Z, Godino J, Multhaup M, Chan DKC, Au Yeung SL, Luo S, Chung BHY, Griffin S, Kim Y. Effects of Communicating Genetic Risk of Type 2 Diabetes and Wearable Technologies on Behavioral Outcomes in East Asians: Statistical Analysis Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Nov 5;14:e65012. doi: 10.2196/65012. PMID 41191904
- [Derived] Kim Y, Godino JG, Cheung FLT, Multhaup M, Chan DKCKC, Chen Z, Ho HHS, Tse THT, Au Yeung SLR, Lou S, Zhang JH, Wang M, Chung B, Griffin S. Effect of communicating genetic risk of type 2 diabetes and wearable technologies on wearable device-measured behavioural outcomes in East Asians: protocol of a randomised controlled trial. BMJ Open. 2024 Dec 4;14(12):e082635. doi: 10.1136/bmjopen-2023-082635. PMID 39632119